CLINICAL TRIAL: NCT04307121
Title: Association of Constipation Inflammatory and Microbial Translocation Markers as Well as Markers of Microbial Translocation Including Endotoxin and Its Antibodies
Brief Title: Association of Constipation Inflammatory and Microbial Translocation Markers
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 108058
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Constipation; Inflammation
Keywords: constipation; microbial translocation; inflammatory markers
MeSH Terms: conditions — Constipation; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Growing evidences showed that patients with chronic constipation accompanied with intestinal dysbiosis. Gut dysbiosis is a harbinger of chronic inflammation, yet the underlying basis is unclear. Plasma level of microbial translocation is a marker of mucosal permeability. Increased mucosal permeability ignites elevated microbial translocation and is a source of systemic immune activation in CKD patients. The passage of microbial components from the gastrointestinal tract into the systemic circulation may be an important contributor to the chronic inflammatory process and subsequent atherosclerosis development. We plan to determine the association constipation with biomarkers of inflammation such monocyte activation and associated cytokines as well as markers of microbial translocation including endotoxin and its antibodies, intestinal barrier proteins of 200 hemodialysis patients.

DETAILED DESCRIPTION:
Study Design and Population

Patients and methods 2.1. Patient selection Two hundred hemodialysis patients are recruited. Functional constipation will be diagnosed according to the Rome IV criteria. Organic lesions of the abdominal cavity and the pelvic floor are excluded in all patients by endoscopic (sigmoidoscopy, colonoscopy, gastroduodenoscopy), radiologic and ultrasonographic evaluation.

This study will be carried out in accordance with the Declaration of Helsinki as revised in 2008. All patients will give written informed consent to participate in the study. All patients in the renal division of Tungs Taichung Metroharbour Hospital were prospectively and consecutively included. The inclusion criteria are

1. Hemodialysis for more than 3 months
2. Age older than 20 years old

The exclusion criteria are a history of chronic inflammatory disease, the presence of current infection, collagen vascular disease or immuno-modulatory or immuno-suppressive treatment.

Measurements of inflammatory cytokines, etotaxin-1, and amyloid A

The plasma levels of MCP-1, IL-6, CRP, IL-17A and calprotectin are tested by commercially available human ELISA kit respectively, according to the manufacturer's instruction. Human serum eotaxin1 levels are determined using a commercial ELISA kit (R&D systems, Minneapolis, MN, USA) according to the manufacturer's protocol. The commercially available ELISA procedure is used to measure serum amyloid A concentration in serum,

Endotoxin and Endotoxin Ig M as well as IgG core antibody

Endotoxin is measured in serum by Limulus Amebocyte Lysate QCL-1000 from Lonza (catalogue # 50-647U)(EU/ml). Serum or plasma samples are diluted at 1∶5 ratio with LAL reagent water. Endotoxin IgG core antibodies are measured in plasma using an ELISA kit from Cell Sciences Inc (catalogue # HK504). Units are expressed as GMU/ml which are IgG standard median units based on medians of ranges of 1000 healthy adults by the manufacturer.

Determination of CD14 and CD16 Mononuclear Phenotype

Peripheral blood will be collected by venipuncture using ethylenedi- aminetetraacetic acid (EDTA) as an anticoagulant. For cytometric analysis, monoclonal antibodies against CD14 (fluorescein isothiocyanate (FITC) conjugated; clone RMO52; Beckman Coulter, Miami, FL, USA), CD16 (phycoerythrin (PE) conjugated; clone 3G8; Beckman Coulter, Miami, FL, USA), CD45 (phycoerythrin cyanin-5 (PC5); clone J33; Beckman Coulter, Miami, FL, USA), and CD56 (clone IM2073; Beckman Coulter, Miami, FL, USA) are used. Briefly, 100 l of the whole blood is stained with saturating amounts of the above mentioned monoclonal antibodies and corresponding isotype controls. After incubation for 15 min at room temperature in the dark according to the manufacturer's recommendations, OptiLyse C (Beckman Coulter, Miami, FL) is added to lyse RBC and the samples are fixed. Fixed cells are analyzed by flow cytometry within 6 hours.

Determination of leukocyte and monocyte subset distribution is performed using a FC500-Cytometer (Beckman Coulter), and CXP analysis software (version 2.2) is used (Schroers et al., 2005). Monocytes are identified as CD45 positive and CD56 negative cells exhibiting a specific forward and sideward scatter profile. Monocytes are then gated in an SSC/CD dot plot, identifying monocytes as CD86 cells with monocyte scatter properties. Subsets of CD14 monocytes with and without CD16 are defined according to the surface expression pattern of the lipopolysaccharide receptor CD14 and the CD16 (Fcgamma receptor III). One million cells are analyzed from each sample, and the percentage of CD16 positive mononuclear cells (CD14+/CD16+ and CD14++/CD16+) and the number of cells out of the total monocytes are compared using fluorescent microbeads (Flow-Count, Beckman Coulter). The CD86 antibody (clone HA5.2B7; Beckman Coulter, Miami, FL, USA) is used in this study.

sCD14, LBP, zonulin and I-FABP assays

LBP and sCD14 markers are used to monitor the microbial translocation while Zonulin and I-FABP are measured to explore intestinal permeability: LBP plasma levels are measured using Enzyme Immunoassay for Quantification of free human LBP ELISA kit, according to the manufacturer's recommendations. Dilution factor is 1:800. Plasma level of sCD14 is measured using Human sCD14 kit, according to the manufacturer's specifications. Dilution factor is 1:200. Zonulin serum levels are measured using Human zonulin ELISA kit. I-FABP plasma levels are measured by ELISA kit according to the manufacturer's recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis for more than 3 months and Age older than 20 years old

Exclusion Criteria:

* he exclusion criteria are a history of chronic inflammatory disease, the presence of current infection, collagen vascular disease or immuno-modulatory or immuno-suppressive treatment.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis (HD) patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Microbial Translocation Markers | 1 years
  Plasma level of microbial translocation is a marker of mucosal permeability. Increased mucosal permeability ignites elevated microbial translocation and is a source of systemic immune activation in CKD patients. microbial translocation including endotoxin and its antibodies, intestinal barrier proteins

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan